CLINICAL TRIAL: NCT00000458
Title: Sertraline and Cognitive Therapy in Depressed Alcoholics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAMOA10476
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: Alcoholism; Depression
MeSH Terms: conditions — Alcoholism; Depression | interventions — Sertraline; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: sertraline (Zoloft)
Behavioral: cognitive behavior therapy

SUMMARY:
This study will assess whether individuals treated with sertraline (Zoloft) and cognitive behavior therapy will experience improvement with their depression and consume less alcohol than individuals treated with a placebo and cognitive behavior therapy. This is a 12-week, random assignment, placebo-controlled, double-blind study with followup assessments 1 and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for major depressive episode.
* Meets criteria for alcohol abuse or dependence thirty days prior to entering the study.
* Has had no more than one previous inpatient medical detoxification.
* Able to maintain sobriety for ten days.
* Able to read and understand questionnaires and informed consent.
* Lives within 50 miles of the study site, has a stable living situation, and a reliable source of collateral reporting.

Exclusion Criteria:

* Meets criteria for any other psychoactive substance dependence other than nicotine.
* Any psychoactive substance abuse (other than nicotine or marijuana) within 30 days before beginning of study.
* Meets criteria for other psychiatric disorders including: panic disorder, obsessive-compulsive disorder, bipolar affective disorder, cyclothymia, schizophrenia, any organic mental disorder, eating disorder, dissociative disorder, or post-traumatic stress disorder.
* Has evidence of treatment resistant depression defined as more than one previous treatment episode for depression, which can include hospitalization and/or one course of antidepressant medication.
* Patients may not have been prescribed a specific serotonergic medication within the month prior to study and may not have taken any antidepressant or antipsychotic within the two weeks prior to study.
* Current use of disulfiram (Antabuse) or anti-seizure medications.
* Clinically significant medical problems: cardiovascular, renal, gastrointestinal, or endocrine problems that would limit participation or limit medication ingestion.
* Hepatocellular disease.
* Females who are pregnant, nursing, or not using a reliable form of birth control.
* Current charges pending for violent crime (excluding DUI related offenses).
* Previous adverse experience with a serotonin reuptake inhibitor.
* Current homicidal or suicidal ideation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States